CLINICAL TRIAL: NCT02860182
Title: Mechanical Characterization of Ascending Aorta in Patients With Acute Type A Dissection and in Healthy Control Group Combined to Structural and Ultrastructural Analysis of Aortic Tissue
Brief Title: Mechanical Characterization of Ascending Aorta in Patients With and Without Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-08
Record Dates: First submitted 2016-07-29; First posted 2016-08-09 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Acute Type A Dissection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- experimental: patients with acute type A dissection
  Interventions: Other: measure the elastic properties of aortic wall
- control: patients without any pathology of the ascending aorta, but having the same characteristics as the sick patients, in terms of age and vascular risk factors including high blood pressure
  Interventions: Other: measure the elastic properties of aortic wall

INTERVENTIONS:
Other: measure the elastic properties of aortic wall

SUMMARY:
Acute type A aortic dissection is a frequent (3 cases per 100 000 people per year) and severe (spontaneous mortality 70%), needing an emergency surgical treatment. Surgical outcomes have improved with the development of surgical techniques, but the postoperative mortality remains high (15-30% at 30 days). Endovascular approach with the deployment of endoprosthesis sealing the proximal intimal tear is an attractive minimally invasive technique, which can represent an alternative to surgical repair especially in high risk patients.

DETAILED DESCRIPTION:
Objectives: this study aims to characterize mechanical properties of ascending aorta (AA) in patients, with and without aortic dissection.

Materials and methods : comprised an in vivo and ex vivo studies performed in 2 groups of patients : (1) patients admitted for acute type A dissection and treated with surgical procedure ; (2) healthy control group selected among patients without any ascending aorta pathology and who underwent transoesophageal echocardiography for various indications.

In vivo study : Strain, distensibility, stiffness index and pressure strain elastic modulus (Ep) were calculated from aortic diameter variation in response to pressure variation. Aortic diameters were measured using transoesophageal echocardiography.

Ex vivo study : biaxial tensile testing were performed on aortic wall samples. Dissected aortic samples were collected from patients who underwent surgical repair and healthy samples from unused donors hearts and lungs. Mechanical characterization was combined to a histological and microstructural analysis of aortic wall. The latter was conducted using multiphoton microscopy to visualize elastin and collagen fibers.

Results :

In vivo study: 22 patients in healthy control group and 13 patients in dissection group were prospectively investigated.

In vitro study : Biaxial testing was performed on 4 samples of dissected aorta and 6 samples of non dissected aorta. Anisotropic and non linear behavior of aortic tissue was shown in the 2 types of samples. Dissected tissue were stiffer than the intimal flap which was in turn stiffer than non dissected tissue.

Histological data showed that in dissection group global elastin density was lower than in control. Microstructural analysis in dissection specimens revealed a higher collagen signal in the media mainly in circumferential plane, contrasting with a roughly similar intensity between the two planes in control. This higher signal reflects higher collagen fiber density and/or thicker fibers in this tunica.

Conclusion : Both in vivo and in vitro data revealed that dissected aorta was stiffer than healthy ascending aorta. These findings has consequences on the choice of futur devices dedicated to AA

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 85 years
* The information given search,
* Aortic dissection evolving for less than 15 days confirmed

Exclusion Criteria:

* the acute aortic dissections against-indicated for aortic surgery (patient age, stroke or multiple organ failure)
* Iatrogenic dissections,
* Dissections related to congenital or hereditary disorder (abnormal connective tissue) or those occurring in subjects with a bicuspid aortic valve,
* Intramural hematomas type A,
* Patients under guardianship or trusteeship deprived of liberty.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ascending aorta dissection
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
measure the elastic properties of aortic wall | one day
  The distensibility, aortic strain will be measured as a function of changes of aortic diameter and pulse pressure.
Measurement of aortic diameters | one day
  The measurement will be done by transesophageal echocardiography simultaneously to the cuff brachial artery pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France